CLINICAL TRIAL: NCT04825678
Title: Phase 4, Open-label Study to Evaluate Treatment Satisfaction With Erenumab in Patients With Migraine
Brief Title: A Study to Evaluate Treatment Satisfaction With Erenumab in Participants With Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20190389
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Migraine
Keywords: Migraine; Chronic Migraine; Episodic Migraine; Erenumab
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erenumab (Experimental)
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Administered as a subcutaneous injection via the SureClick® Autoinjector Pen (AI/Pen).
  Other Names: AMG 334

SUMMARY:
The main purpose of this study is to evaluate the effect of erenumab on medication-specific treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Participant has provided informed consent
* History of migraine (with or without aura) for ≥ 12 months before screening
* ≥ 4 migraine days per month on average across the 3 months prior to screening
* Treatment with 1 oral migraine preventive medication and/or concomitant use of OnabotulinumtoxinA injections for migraine prevention.
* Participant reports to their provider intolerance or insufficient response with their current preventative treatment

Exclusion Criteria:

* History of cluster headache or hemiplegic migraine headache
* Unable to differentiate migraine from other headaches
* Evidence of substance-related disorders
* Active chronic pain syndromes (eg, fibromyalgia and chronic pelvic pain)
* No therapeutic response with > 3 migraine preventive medication categories
* Used a prohibited medication, device, or procedure
* Other clinically significant disorder, condition, or disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (42):
- United States (42):
  - Rehabilitation and Neurological Services LLC, Huntsville, Alabama
  - Elite Clinical Studies LLC, Phoenix, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - The Neurology Group, Pomona, California
  - Mountain Neurological Research Center, Basalt, Colorado
  - Mindscapes Counseling, LLC, Norwich, Connecticut
  - Reliable Clinical Research, LLC, Hialeah, Florida
  - Homestead Associates In Research Inc, Homestead, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - The Community Research of South Florida, Miami Lakes, Florida
  - Research Institute of Orlando, Orlando, Florida
  - Pas Research, Tampa, Florida
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Chicago Headache Center and Research Institute, Chicago, Illinois
  - College Park Family Care Center, Overland Park, Kansas
  - Family HealthCare, Germantown, Maryland
  - Neurology Center of New England, Foxborough, Massachusetts
  - ActivMed Practices and Research, LLC, Lowell, Massachusetts
  - Memorial Healthcare Foundation, Owosso, Michigan
  - SRI International, Plymouth, Michigan
  - Citizens Memorial Healthcare, Bolivar, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Psych Care Consultants, St Louis, Missouri
  - Albuquerque Clinical Trials Inc, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Dent Neurosciences Research Center, Amherst, New York
  - Northwell Health Physician Partners Neuroscience Institute at Great Neck, Great Neck, New York
  - Island Neurological Associates, Plainview, New York
  - Nuvance Health Medical Practice Primary Care Division of Neurology, Poughkeepsie, New York
  - Montefiore Medical Center, The Bronx, New York
  - Asheville Neurology Specialists PA, Asheville, North Carolina
  - Onsite Clinical Solutions LLC, Charlotte, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Saint Lukes Neurology Associates, Bethlehem, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Premier Neurology, Greer, South Carolina
  - Tri-State Mountain Neurology Associates, Johnson City, Tennessee
  - Pearland Neurology Services PLLC, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Houston Neurology Associates, Sugar Land, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - Vaught Neurological Services, Crab Orchard, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 33 centers in the United States (US) from June 2021 to September 2023.
Pre-assignment Details: This study enrolled participants with episodic migraine (EM) or chronic migraine (CM) in an approximately 1:1 ratio. The study comprised of a combined screening/baseline period and a 24-week open-label treatment period.
Groups:
- Erenumab QM: EM: Participants with EM were administered erenumab QM subcutaneously (SC). EM was defined as < 15 headache days a month over the last 3 months, which on some days was migraine but did not fulfil International Headache Society (IHS) International Classification of Headache Disorders (ICHD) Classification III criteria for CM per participant self-report and investigator assessment.
  All participants started on a 70 mg dose of erenumab at Day 1 with provider discretion for dose optimization (either 70 mg or 140 mg), which was recommended to be completed by Week 12. All participants were required to enter the study on 1 standard of care preventive medication for their migraine, whose dose then could be adjusted by the investigator's discretion and were stable by Week 12.
  No dose comparisons were pre-specified.
- Erenumab QM: CM: Participants with CM were administered erenumab QM SC. CM was defined as ≥ 15 headache days a month of which ≥ 8 headache days met criteria as migraine days per participant self-report and investigator assessment.
  All participants started on a 70 mg dose of erenumab at Day 1 with provider discretion for dose optimization (either 70 mg or 140 mg), which was recommended to be completed by Week 12. All participants were required to enter the study on 1 standard of care preventive medication for their migraine, whose dose then could be adjusted by the investigator's discretion and were stable by Week 12.
  No dose comparisons were pre-specified.
Period: Overall Study
Arm/Group | Erenumab QM: EM | Erenumab QM: CM
Started | 53 | 187
Received Investigational Product | 52 | 186
Received Erenumab QM 70 mg (Participants who remained on 70 mg and did not receive any 140 mg dose) | 32 | 124
Received Erenumab QM 140 mg (Participants who increased dose to 140 mg) | 20 | 62
Continued Standard of Care (SoC) (Participants who continued SoC migraine prevention therapy throughout the study) | 41 | 171
Discontinued SoC (Participants who discontinued SoC migraine prevention therapy during the study) | 12 | 16
Completed | 40 | 170
Not Completed | 13 | 17
Not completed — Decision by Sponsor | 2 | 3
Not completed — Withdrawal of Consent From Study | 7 | 9
Not completed — Lost to Follow-up | 3 | 4
Not completed — Never Received Investigational Product | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): consisted of all participants enrolled in the study.
Groups:
- Erenumab QM: EM: Participants with EM were administered erenumab QM SC. EM was defined as < 15 headache days a month over the last 3 months, which on some days was migraine but did not fulfil IHS Classification ICHD III criteria for CM per participant self-report and investigator assessment.
  All participants started on a 70 mg dose of erenumab at Day 1 with provider discretion for dose optimization (either 70 mg or 140 mg), which was recommended to be completed by Week 12. All participants were required to enter the study on 1 standard of care preventive medication for their migraine, whose dose then could be adjusted by the investigator's discretion and were stable by Week 12.
  No dose comparisons were pre-specified.
- Total: Total of all reporting groups
Arm/Group | Erenumab QM: EM | Erenumab QM: CM | Total
Number analyzed (Participants) | 53 | 187 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (12.7) | 47.0 (14.1) | 46.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 169 | 212
  Male | 10 | 18 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 103 | 116
  Not Hispanic or Latino | 40 | 84 | 124
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Black or African American | 7 | 20 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 43 | 162 | 205
  Other | 2 | 3 | 5
  Multiple | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Treatment Satisfaction Questionnaire for Medication (TSQM) Overall Satisfaction Scale Score at Week 24 by SoC
Description: The TSQM version 1.4 is a 14-item instrument designed to measure important dimensions of participants' experiences with their medication. It has 4 domains: effectiveness, side effects, convenience, and overall satisfaction. Overall satisfaction scores could range from 0 to 100, with higher scores indicating greater satisfaction. A positive change from Baseline represents an increase in overall medication satisfaction.
  Worst postbaseline value observed up to erenumab discontinuation was used for participants who discontinued erenumab due to lack of efficacy or adverse event; missing value used for participants who discontinued erenumab due to other reasons.
Time Frame: Baseline and Week 24
Population: Efficacy Analysis Set (EAS): consists of a subset of participants from FAS who receive at least 1 dose of investigational product. Data presented by SoC migraine preventive treatment, as pre-specified in SAP section 9.5. Only participants with available data were included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Erenumab QM: Continued SoC: Participants with EM and CM who were administered erenumab QM SC and continued SoC migraine prevention therapy throughout the study.
  All participants started on a 70 mg dose of erenumab at Day 1 with provider discretion for dose optimization (either 70 mg or 140 mg), which was recommended to be completed by Week 12. All participants were required to enter the study on 1 standard of care preventive medication for their migraine, whose dose then could be adjusted by the investigator's discretion and were stable by Week 12.
  No dose comparisons were pre-specified.
- Erenumab QM: Discontinued SoC: Participants with EM and CM who were administered erenumab QM SC and discontinued SoC migraine prevention therapy at any point throughout the study.
  All participants started on a 70 mg dose of erenumab at Day 1 with provider discretion for dose optimization (either 70 mg or 140 mg), which was recommended to be completed by Week 12. All participants were required to enter the study on 1 standard of care preventive medication for their migraine, whose dose then could be adjusted by the investigator's discretion and were stable by Week 12.
  No dose comparisons were pre-specified.
Arm/Group | Erenumab QM: Continued SoC | Erenumab QM: Discontinued SoC
Number analyzed (Participants) | 184 | 14
Score on a scale | 42.33 (32.48) | 34.42 (57.66)
Statistical Analysis 1: Comparison: Erenumab QM: Continued SoC; Adjusted analysis utilizes a generalized linear mixed model which includes Baseline TSQM overall satisfaction scale score, visit, the prevailing erenumab dose from Week 12 onwards, observed Baseline monthly migraine days (MMD), and selected Baseline characteristics as covariates and assumes a first-order auto regression covariance structure; Test type: Other; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; Least squares mean (LSM) = 40.72, 95% CI 2-sided [36.05 to 45.39], Standard Error of Mean 2.37
Statistical Analysis 2: Comparison: Erenumab QM: Discontinued SoC; Adjusted analysis utilizes a generalized linear mixed model which includes Baseline TSQM overall satisfaction scale score, visit, the prevailing erenumab dose from Week 12 onwards, observed Baseline MMD, and selected Baseline characteristics as covariates and assumes a first-order auto regression covariance structure; Test type: Other; p = 0.058, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = 30.84, 95% CI 2-sided [-1.30 to 62.98], Standard Error of Mean 14.53

2. Primary Outcome: Mean Change From Baseline in the Treatment Satisfaction Questionnaire for Medication (TSQM) Overall Satisfaction Scale Score at Week 24 by Migraine Type
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: EAS: consists of a subset of participants from FAS who receive at least 1 dose of investigational product. Data presented by migraine type, as pre-specified in SAP section 9.5. Only participants with available data were included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Erenumab QM: EM | Erenumab QM: CM
Number analyzed (Participants) | 38 | 160
Score on a scale | 34.76 (44.00) | 43.44 (32.03)
Statistical Analysis 1: Comparison: Erenumab QM: EM; [analysis description as in outcome 1, analysis 2]; Test type: Other; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = 37.87, 95% CI 2-sided [28.62 to 47.12], Standard Error of Mean 4.62
Statistical Analysis 2: Comparison: Erenumab QM: CM; [analysis description as in outcome 1, analysis 2]; Test type: Other; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = 43.25, 95% CI 2-sided [38.06 to 48.44], Standard Error of Mean 2.63

3. Secondary Outcome: Observed Data: Percentage of Participants Achieving Overall Satisfaction at Week 24 by SoC
Description: Overall satisfaction is defined as the percentage of participants reporting of satisfied, very satisfied, or extremely satisfied on item 14 of the TSQM version 1.4. Item 14 of the TSQM measures global satisfaction on a 7 point rating scale where 1 indicates least satisfaction and 7 indicates most satisfaction.
  Summary statistics using observed data (after intercurrent event handling) presented. The 95% confidence interval (CI) is for the percentage of responders and was calculated using the Clopper-Pearson method.
Time Frame: Week 24
Population: EAS: consists of a subset of participants from FAS who receive at least 1 dose of investigational product. Data presented by SoC migraine preventive treatment, as pre-specified in SAP section 9.5. Only participants with available data were included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Erenumab QM: Continued SoC | Erenumab QM: Discontinued SoC
Number analyzed (Participants) | 188 | 15
Percentage of participants | 91.0 [85.92 to 94.64] | 66.7 [38.38 to 88.18]

4. Secondary Outcome: GLIMMIX Model Data: Percentage of Participants Achieving Overall Satisfaction at Week 24 by SoC
Description: Overall satisfaction is defined as the percentage of participants reporting of satisfied, very satisfied, or extremely satisfied on item 14 of the TSQM version 1.4. Item 14 of the TSQM measures global satisfaction on a 7 point rating scale where 1 indicates least satisfaction and 7 indicates most satisfaction.
  The estimated percentage and CI presented were obtained from a generalized linear mixed model with a logit link which includes Baseline achievement of overall satisfaction, visit, observed Baseline MMD, and selected Baseline characteristics as covariates and assumes a first-order auto regression covariance structure. The model includes data from all visits during treatment period. The 95% CI is for the percentage of responders and was calculated using the Clopper-Pearson method.
Time Frame: Baseline up to Week 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Estimated percentage of participants
Arm/Group | Erenumab QM: Continued SoC | Erenumab QM: Discontinued SoC
Number analyzed (Participants) | 197 | 15
Estimated percentage of participants | 91.8 [81.64 to 96.54] | NA [NA to NA] — Due to limited number of participants, the GLIMMIX model did not converge.

5. Secondary Outcome: Observed Data: Percentage of Participants Achieving Overall Satisfaction at Week 24 by Migraine Type
Description: Overall satisfaction is defined as the percentage of participants reporting of satisfied, very satisfied, or extremely satisfied on item 14 of the TSQM version 1.4. Item 14 of the TSQM measures global satisfaction on a 7 point rating scale where 1 indicates least satisfaction and 7 indicates most satisfaction.
  Summary statistics using observed data (after intercurrent event handling) presented. The 95% CI is for the percentage of responders and was calculated using the Clopper-Pearson method.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Erenumab QM: EM | Erenumab QM: CM
Number analyzed (Participants) | 41 | 162
Percentage of participants | 75.6 [59.70 to 87.64] | 92.6 [87.42 to 96.11]

6. Secondary Outcome: GLIMMIX Model Data: Percentage of Participants Achieving Overall Satisfaction at Week 24 by Migraine Type
Description: as for outcome 4
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Estimated percentage of participants
Arm/Group | Erenumab QM: EM | Erenumab QM: CM
Number analyzed (Participants) | 45 | 167
Estimated percentage of participants | 76.2 [58.50 to 87.90] | 93.2 [84.16 to 97.23]

7. Secondary Outcome: Observed Data: Percentage of Participants Reporting Improvement in the Migraine Global Impression Item (mGI-I) at Week 24 by SoC
Description: Improvement is defined as the percentage of participants reporting of much improved or a little improved on the mGI-I. The mGI-I is a single item instrument designed to measure improvement/worsening in migraine. The 3 versions of the instrument include the perspective of study participants, treating clinicians, and key family members measured on the following scale: much improved; a little improved; no change; a little worse; or much worse. The recall period is the past 7 days.
  Summary statistics using observed data (after intercurrent event handling) presented. The 95% CI is for the percentage of responders and was calculated using the Clopper-Pearson method.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Erenumab QM: Continued SoC | Erenumab QM: Discontinued SoC
Number analyzed (Participants) | 189 | 13
Percentage of participants
  Participant Global Impression: number analyzed (Participants) | 151 | 12
  Participant Global Impression | 94.0 [88.99 to 97.24] | 83.3 [51.59 to 97.91]
  Treating Clinician's Global Impression | 93.7 [89.17 to 96.68] | 84.6 [54.55 to 98.08]
  Key Family Member's Impression: number analyzed (Participants) | 83 | 4
  Key Family Member's Impression | 92.8 [84.93 to 97.30] | 100.0 [39.76 to 100.0]

8. Secondary Outcome: GLIMMIX Model Data: Percentage of Participants Reporting Improvement in the mGI-I at Week 24 by SoC
Description: Improvement is defined as the percentage of participants reporting of much improved or a little improved on the mGI-I. The mGI-I is a single item instrument designed to measure improvement/worsening in migraine. The 3 versions of the instrument include the perspective of study participants, treating clinicians, and key family members measured on the following scale: much improved; a little improved; no change; a little worse; or much worse. The recall period is the past 7 days.
  The estimated percentage and CI presented were obtained from a generalized linear mixed model with a logit link which includes visit, observed Baseline MMD, and selected Baseline characteristics as covariates and assumes a first-order auto regression covariance structure. The model includes data from all visits during treatment period. The 95% CI is for the percentage of responders and was calculated using the Clopper-Pearson method.
Time Frame: Baseline up to Week 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Estimated percentage of participants
Arm/Group | Erenumab QM: Continued SoC | Erenumab QM: Discontinued SoC
Number analyzed (Participants) | 202 | 13
Estimated percentage of participants
  Participant Global Impression: number analyzed (Participants) | 174 | 12
  Participant Global Impression | 94.6 [87.42 to 97.82] | NA [NA to NA] — Due to limited number of participants, the GLIMMIX model did not converge.
  Treating Clinician's Global Impression | 90.9 [82.71 to 95.46] | NA [NA to NA] — Due to limited number of participants, the GLIMMIX model did not converge.
  Key Family Member's Impression: number analyzed (Participants) | 114 | 5
  Key Family Member's Impression | 92.6 [81.09 to 97.37] | NA [NA to NA] — Due to limited number of participants, the GLIMMIX model did not converge.

9. Secondary Outcome: Observed Data: Percentage of Participants Reporting Improvement in the mGI-I at Week 24 by Migraine Type
Description: as for outcome 7
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Erenumab QM: EM | Erenumab QM: CM
Number analyzed (Participants) | 40 | 162
Percentage of participants
  Participant Global Impression: number analyzed (Participants) | 31 | 132
  Participant Global Impression | 83.9 [66.27 to 94.55] | 95.5 [90.37 to 98.31]
  Treating Clinician's Global Impression | 87.5 [73.20 to 95.81] | 94.4 [89.72 to 97.43]
  Key Family Member's Impression: number analyzed (Participants) | 14 | 73
  Key Family Member's Impression | 85.7 [57.19 to 98.22] | 94.5 [86.56 to 98.49]

10. Secondary Outcome: GLIMMIX Model Data: Percentage of Participants Reporting Improvement in the mGI-I at Week 24 by Migraine Type
Description: as for outcome 8
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Estimated percentage of participants
Arm/Group | Erenumab QM: EM | Erenumab QM: CM
Number analyzed (Participants) | 46 | 169
Estimated percentage of participants
  Participant Global Impression: number analyzed (Participants) | 36 | 150
  Participant Global Impression | NA [NA to NA] — Due to limited number of participants, the GLIMMIX model did not converge. | 95.5 [88.89 to 98.23]
  Treating Clinician's Global Impression | 87.3 [65.28 to 96.15] | 94.5 [85.74 to 98.02]
  Key Family Member's Impression: number analyzed (Participants) | 18 | 101
  Key Family Member's Impression | NA [NA to NA] — Due to limited number of participants, the GLIMMIX model did not converge. | NA [NA to NA] — Due to limited number of participants, the GLIMMIX model did not converge.

11. Secondary Outcome: Mean Change From Baseline in Domain Scores as Measured by the Migraine Functional Impact Questionnaire (MFIQ) at Week 24 by SoC
Description: The MFIQ version 2.0 is a self-administered 26-item instrument measuring the impact of migraine on broader functioning including 4 domains: Impact on Physical Functioning, Impact on Usual Activities, Impact on Social Functioning, and Impact on Emotional Functioning. In addition, there is 1 stand-alone global item assessing the overall impact on usual activities. Participants respond to each item using a 5-point scale assigned scores from 1 to 5, with 5 representing the greatest burden. Each domain score was calculated as the sum of the item responses (i.e., raw score) and rescaled to a 0-100 scale, with higher scores representing greater burden. A negative change from baseline represents a reduction in burden. The recall period is the past 7 days.
  Summary statistics using observed data (after intercurrent event handling) presented.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Erenumab QM: Continued SoC | Erenumab QM: Discontinued SoC
Number analyzed (Participants) | 185 | 13
Score on a scale
  Physical Function Domain | -46.29 (26.70) | -49.04 (30.20)
  Usual Activities Domain | -44.83 (25.08) | -45.00 (27.86)
  Social Function Domain | -45.87 (27.62) | -46.15 (30.63)
  Emotional Function Domain | -47.54 (29.33) | -57.31 (31.73)
Statistical Analysis 1: Comparison: Erenumab QM: Continued SoC; Continued SoC: Physical Function Domain; Test type: Other — Adjusted analysis utilizes a generalized linear mixed model which includes Baseline function domain score, visit, the prevailing erenumab dose from Week 12 onwards, observed Baseline MMD, and selected Baseline characteristics as covariates and assumes a first-order auto regression covariance structure; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -44.90, 95% CI 2-sided [-49.39 to -40.41], Standard Error of Mean 2.28
Statistical Analysis 2: Comparison: Erenumab QM: Discontinued SoC; Discontinued SoC: Physical Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -54.15, 95% CI 2-sided [-73.43 to -34.86], Standard Error of Mean 8.43
Statistical Analysis 3: Comparison: Erenumab QM: Continued SoC; Continued SoC: Usual Activities Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from baseline at Week 24 to zero; LSM = -44.35, 95% CI 2-sided [-48.26 to -40.44], Standard Error of Mean 1.99
Statistical Analysis 4: Comparison: Erenumab QM: Discontinued SoC; Discontinued SoC: Usual Activities Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -43.80, 95% CI 2-sided [-53.51 to -34.08], Standard Error of Mean 4.47
Statistical Analysis 5: Comparison: Erenumab QM: Continued SoC; Continued SoC: Social Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -44.39, 95% CI 2-sided [-48.65 to -40.14], Standard Error of Mean 2.16
Statistical Analysis 6: Comparison: Erenumab QM: Discontinued SoC; Discontinued SoC: Social Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -45.03, 95% CI 2-sided [-60.28 to -29.79], Standard Error of Mean 6.97
Statistical Analysis 7: Comparison: Erenumab QM: Continued SoC; Continued SoC: Emotional Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -45.50, 95% CI 2-sided [-50.29 to -40.70], Standard Error of Mean 2.44
Statistical Analysis 8: Comparison: Erenumab QM: Discontinued SoC; Discontinued SoC: Emotional Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -60.06, 95% CI 2-sided [-85.16 to -34.96], Standard Error of Mean 10.98

12. Secondary Outcome: Mean Change From Baseline in Domain Scores as Measured by the MFIQ at Week 24 by Migraine Type
Description: as for outcome 11
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Erenumab QM: EM | Erenumab QM: CM
Number analyzed (Participants) | 38 | 160
Score on a scale
  Physical Function Domain | -29.84 (26.08) | -50.42 (25.58)
  Usual Activities Domain | -32.22 (26.47) | -47.84 (24.00)
  Social Function Domain | -32.99 (30.50) | -48.95 (26.23)
  Emotional Function Domain | -37.50 (34.66) | -50.72 (27.67)
Statistical Analysis 1: Comparison: Erenumab QM: EM; EM: Physical Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -34.38, 95% CI 2-sided [-41.72 to -27.03], Standard Error of Mean 3.69
Statistical Analysis 2: Comparison: Erenumab QM: CM; CM: Physical Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -49.56, 95% CI 2-sided [-54.44 to -44.69], Standard Error of Mean 2.48
Statistical Analysis 3: Comparison: Erenumab QM: EM; EM: Usual Activities Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from baseline at Week 24 to zero; LSM = -35.76, 95% CI 2-sided [-41.47 to -30.06], Standard Error of Mean 2.88
Statistical Analysis 4: Comparison: Erenumab QM: CM; CM: Usual Activities Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -46.70, 95% CI 2-sided [-51.10 to -42.29], Standard Error of Mean 2.23
Statistical Analysis 5: Comparison: Erenumab QM: EM; EM: Social Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -36.42, 95% CI 2-sided [-42.89 to -29.96], Standard Error of Mean 3.26
Statistical Analysis 6: Comparison: Erenumab QM: CM; CM: Social Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -46.73, 95% CI 2-sided [-51.49 to -41.98], Standard Error of Mean 2.41
Statistical Analysis 7: Comparison: Erenumab QM: EM; EM: Emotional Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -41.44, 95% CI 2-sided [-49.47 to -33.40], Standard Error of Mean 4.04
Statistical Analysis 8: Comparison: Erenumab QM: CM; CM: Emotional Function Domain; Test type: Other — [test comment as in outcome 11, analysis 1]; p < 0.001, Mixed Models Analysis — P-value is nominal to compare the mean change from Baseline at Week 24 to zero; LSM = -47.67, 95% CI 2-sided [-52.95 to -42.39], Standard Error of Mean 2.68

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. Data presented by SoC migraine preventive treatment, as pre-specified in SAP section 9.6.
Groups:
- Erenumab QM: Total: All participants with EM and CM who were administered erenumab QM SC.
  All participants started on a 70 mg dose of erenumab at Day 1 with provider discretion for dose optimization (either 70 mg or 140 mg), which was recommended to be completed by Week 12. All participants were required to enter the study on 1 standard of care preventive medication for their migraine, whose dose then could be adjusted by the investigator's discretion and were stable by Week 12.
  No dose comparisons were pre-specified.
Arm/Group | Erenumab QM: Continued SoC | Erenumab QM: Discontinued SoC | Erenumab QM: Total
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/28 | 0/240
Serious Adverse Events (participants affected / at risk) | 5/212 | 1/26 | 6/238
Other Adverse Events (participants affected / at risk) | 16/212 | 7/26 | 23/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab QM: Continued SoC (N=212) | Erenumab QM: Discontinued SoC (N=26) | Erenumab QM: Total (N=238)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab QM: Continued SoC (N=212) | Erenumab QM: Discontinued SoC (N=26) | Erenumab QM: Total (N=238)
Constipation (Gastrointestinal disorders) | 10 | 3 | 13
Injection site erythema (General disorders) | 0 | 2 | 2
COVID-19 (Infections and infestations) | 8 | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT04825678/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT04825678/SAP_001.pdf